CLINICAL TRIAL: NCT01067586
Title: Toxicant Exposure Across Brands of Smokeless Tobacco
Brief Title: Novel Determinants and Measures of Smokeless Tobacco Use: Study 1
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009NTUC053; 1R01CA141531 (NIH)
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Smokeless Tobacco Use; Tobacco Dependence
Keywords: Smokeless Tobacco; Biomarkers of tobacco exposure
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, buccal cells and blood will be collected from subjects in this study.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The extent of toxicity varies considerably across different brands of smokeless tobacco (ST) products and data suggest that greater toxicity may result in greater health risks. However, little is known about the actual extent of exposure to toxicants from current smokeless tobacco products and factors that might moderate the extent of this exposure. The goals of this project are to address the following questions:

1. What are the characteristics of the range of smokeless tobacco products in current use and how do these products impact user behavior;
2. What are novel and the best measures of smokeless tobacco use, behavior and exposure; and
3. What are some of the determinants of smokeless tobacco use.

DETAILED DESCRIPTION:
Study 1 is a multi-site descriptive study assessing tobacco toxicants in various smokeless tobacco products and tobacco toxicant exposure found in 600 subjects in three sites: University of MN Twin Cities, Oregon Research Institute in Eugene OR, and at West Virginia University in Morgantown, WV (200 subjects per site). The study will examine the relationship between brands of U.S. smokeless tobacco products that contain different levels of tobacco-specific nitrosamines (TSNAs), other carcinogens and nicotine, and biomarkers of exposure and effects on health (e.g., cardiovascular risk factors). Additionally, the study will examine factors that influence the extent of toxicant exposure and effect besides the levels of toxicants in the product. Subjects will attend an orientation where they will sign a consent form and then return for one clinic visit where they will provide blood (UMN only), urine samples, buccal samples and expectorated chews to be examined for nicotine levels, toxicant exposure and potential for tobacco-related health risks. A subsample of subjects (10 per brand of smokeless tobacco) will be asked for a tin of their unused product for testing (they will be reimbursed for the cost of their tin) and will be asked for three samples of expectorated chews that will be collected, frozen and shipped to the CDC where they will be analyzed for tobacco constituents. Subjects will complete several questionnaires on their tobacco use history, alcohol, diet, physical and mental health. Subjects will also keep a daily diary of their tobacco and alcohol use.

ELIGIBILITY:
Inclusion Criteria:

1. Using a consistent and daily amount of ST for the past year;
2. In good physical health (no unstable medical condition);
3. Stable, good mental health (e.g., no recent unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the DSM-IV criteria).

Exclusion Criteria:

1. Subjects must not be currently using other tobacco or nicotine products.
2. Female subjects cannot be pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokeless tobacco users of 6 brands of tobacco
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2010-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of MN's Tobacco Use Research Center, Minneapolis, Minnesota
  - Oregon Research Institute, Eugene, Oregon
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Daily users of certain smokeless tobacco products who were 18 years or older were recruited in Minneapolis/St. Paul, MN, Eugene, OR and Morgantown, WV via local advertisements. Subjects were recruited from 2/2010 through 5/2012.
Groups:
- Smokeless Tobacco Users: x
Period: Overall Study
Arm/Group | Smokeless Tobacco Users
Started | 359
Completed | 359
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Smokeless Tobacco Users
Number analyzed (Participants) | 359
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 352
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 357
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 331
  More than one race | 10
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 359
History of smoking >100 cigarettes [Count of Participants; unit: Participants] | 350
Age of initiation [Mean (Standard Deviation); unit: years] | 17.7 (8.5)
Duration of use [Mean (Standard Deviation); unit: years] | 13.9 (11.9)
Tins per wek [Mean (Standard Deviation); unit: tins per week] | 3.6 (2.2)
Mean dips per day [Mean (Standard Deviation); unit: Mean dips per day] | 7.0 (3.5)
Mean duration of dip [Mean (Standard Deviation); unit: minutes] | 69.3 (42.0)
Total nicotine equivalents (TNE) [Mean (Standard Deviation); unit: nmol/mg] | 72.8 (70.9)
Total NNAL [Mean (Standard Deviation); unit: pmol/mg creatinine] | 3.29 (3.77)
Total NNN [Mean (Standard Deviation); unit: pmol/mg creatinine] | 0.284 (3.374)

OUTCOME MEASURES:

1. Primary Outcome: Extent of Toxicity: Mean of Median Values of NNK+NNN in 7 Smokeless Tobacco Brands
Description: Two important harmful constituents in smokeless tobacco products are NNN + NNK, µg/g This measure reports the tobacco-specific nitrosamines (TSNA), N'-nitrosonornicotine (NNN), and 4- (methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK) across 7 different smokeless tobacco brands.
Time Frame: Three "usual" dip sized samples were collected from subjects at baseline
Population: Products included samples from Copenhagen (Copenhagen Snuff, Copenhagen Long Cut, Copenhagen Long Cut Straight, Copenhagen Long Cut Wintergreen)
Measure: Mean (Full Range); unit: ug/g
Units Other Than Participants: brand variety
Groups:
- Copenhagen: Products included Copenhagen Snuff, Copenhagen Long Cut, Copenhagen Long Cut Straight, Copenhagen Long Cut Wintergreen
- Skoal: Skoal samples include Skoal Long Cut Straight, Skoal Fine Cut Original, Skoal Long Cut Wintergreen, Skoal Bandits Wintergreen, Skoal Long Cut Mint, Skoal Wintergreen Pouches, Skoal Mint Pouches, Skoal Snus
- Kodiak: Kodiak includes Kodiak Wintergreen, Kodiak Wintergreen Moist Snuff Pouches
- Grizzly: Products include Grizzly Long Cut Straight, Grizzly Strait Pouches, Grizzly Fine Cut Natural, Grizzly Long Cut Mint, Grizzly Mint Pouches, Grizzly Long Cut Wintergreen, Grizzly Wintergreen Pouches
- Red Seal: Product is Red Seal Fine Cut Natural
- Marlboro Snus: Products include Marlboro Snus Original, Marlboro Snus Peppermint, Marlboro Snus Mint, Marlboro Snus Rich
- Camel Snus: Products include Camel Snus Robust, Camel Snus Mellow, Camel Snus Frost, Camel Snus Winterchill
Arm/Group | Copenhagen | Skoal | Kodiak | Grizzly | Red Seal | Marlboro Snus | Camel Snus
Number analyzed (Participants) | 110 | 60 | 26 | 132 | 12 | 5 | 30
Number analyzed (brand variety) | 4 | 9 | 2 | 7 | 1 | 4 | 4
ug/g | 2.4 [1.23 to 3.42] | 2.25 [1.25 to 3.89] | 3.19 [2.97 to 3.40] | 5.51 [3.04 to 14.55] | 2.61 [2.61 to 2.61] | 0.74 [0.64 to 0.78] | 1.73 [1.66 to 1.79]

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed. Outcomes evaluated were on tobacco products, not human participants, so no adverse events were possible.
Groups:
- Smokeless Tobacco Brands: x
Arm/Group | Smokeless Tobacco Brands
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2009-12-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT01067586/Prot_SAP_000.pdf
  • Informed Consent Form (2011-06-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT01067586/ICF_001.pdf